CLINICAL TRIAL: NCT05491824
Title: Bio-Repository of DNA in Stroke: an Epidemiological and Genetic Study
Acronym: BRAINS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Holloway University (Other)
Responsible Party: Principal Investigator, Pankaj Sharma, MD PhD, Professor, Royal Holloway University
Other Study IDs: BRAINS
Record Dates: First submitted 2022-08-02; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Stroke; Stroke, Ischemic; Stroke Hemorrhagic
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke
- Non-stroke

SUMMARY:
The Bio-Repository of DNA in Stroke (BRAINS) recruits all subtypes of stroke as well as controls from two different continents, Europe and Asia. Subjects recruited from the United Kingdom (UK) will include stroke patients of European ancestry as well as British South Asians. Stroke subjects from South Asia will be recruited from India and Sri Lanka. Subjects are also recruited in Qatar. South Asian cases will also have control subjects recruited.

ELIGIBILITY:
Cases

Inclusion Criteria:

* Patients should be aged > 18 years at the time of enrolment.
* Diagnosis of haemorrhagic or ischemic stroke using World Health Organization guidelines confirmed by clinical examination and imaging (CT or MRI).
* All patients with cerebral arteriovascular malformations and aneurysms.
* South Asian or Caucasian ethnic backgrounds.
* Patient or relative written informed consent.

Exclusion Criteria:

* Unable to provide consent themselves or through surrogate.
* Stroke not defined on CT or MRI.

Controls

Inclusion Criteria:

* Patients should be aged > 18 years at the time of enrolment.
* No previous history of stroke.
* able to provide written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients and spouse or age-matched controls will be screened at the participating clinical centres in the United Kingdom (London, Luton, Birmingham, Leeds, Leicester, Airedale, Bradford, Wolverhampton and Blackburn), India (New Delhi and Kerala), Qatar and Sri Lanka (Colombo). Detailed phenotype data will be collected in a specially designed BRAINS data collection form. Stroke will be confirmed with computed tomography or magnetic resonance imaging and subtyped according to the Trial of ORG10172 in Acute Stroke Treatment (TOAST) classification. Baseline clinical and demographic data will also be collected. Blood samples will be collected in EDTA coated plastic serological tubes from all consenting patients and controls by means of a single venepuncture and DNA extracted from peripheral lymphocytes using standard procedure and stored at -20°C. Following genotyping the genetic data will be merged with phenotype data (environmental risk factors, stroke sub-type) for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2005-06-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
DNA repository of highly phenotyped stroke patients | 5 years
Identify novel gene loci associated with different types of stroke | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Sharma, MD PhD, Principal Investigator — Royal Holloway University
Locations (1):
- Imperial College London, London, United Kingdom